CLINICAL TRIAL: NCT06202300
Title: Myocardial and Arterial Phenotype of Coronary Artery Disease (CAD-MAP): A Multicenter Multimodality Imaging & Physiology Registry
Brief Title: Myocardial and Arterial Phenotype of Coronary Artery Disease
Acronym: CAD-MAP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Xiao Wang, Chief Physician, Beijing Anzhen Hospital
Other Study IDs: KS2023013
Record Dates: First submitted 2024-01-01; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Multimodality imaging; Inflammation; Clinical outcome
MeSH Terms: conditions — Coronary Artery Disease; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with high inflammation level: CAD patients undergoing multimodality imaging with high inflammation burden
  Interventions: Other: Inflammation burden
- Patients with low inflammation level: CAD patients undergoing multimodality imaging with low inflammation burden
  Interventions: Other: Inflammation burden

INTERVENTIONS:
Other: Inflammation burden — Coronary artery disease patients undergone multimodality imaging with different level inflammation burden

SUMMARY:
The CAD-MAP (Myocardial and Arterial Phenotype of Coronary Artery Disease) registry is initiated with the goal to describe the cardiac imaging map including epicardial coronary artery, coronary microcirculation and myocardium, and further exploring the prognostic value of multidimensional imaging biomarkers and predictive models in CAD patients.

DETAILED DESCRIPTION:
Despite advances in medical therapy and the greater use of reperfusion therapy, morbidity and mortality following coronary artery disease (CAD) remains substantial, with increase in elder population and the epidemic of metabolic risk factors. The pathophysiological process of CAD involves the pathological changes of myocardium and coronary arteries. Current risk stratification based on traditional risk factors and clinical characteristics cannot reflect the comprehensive effects of risk factors on pathological features, thus providing limited prognostic value in CAD patients.

Invasive and noninvasive cardiovascular imaging techniques including vascular and myocardial imaging can lead to a better understanding of underlying pathological mechanisms of CAD and further improve phenotyping, thus allowing imaging-guided risk stratification and optimizing treatment effects. Coronary computed tomography angiography (CCTA), cardiac magnetic resonance (CMR), and positron emission tomography/computed tomography (PET/CT), which can directly capture coronary and myocardial features, offers a unique tool for the quantification of pathophysiological feature and for better risk stratification of CAD patients.

Current imaging cohorts, including UK Biobank, MESA and PESA, allow for evaluation of atherosclerosis cardiovascular disease. However, these cohorts aimed to evaluate the progression of subclinical atherosclerosis for primary prevention. Moreover, most imaging cohorts of secondary prevention included single imaging modality and few investigated the clinical effect of multimodality imaging-guided treatment in CAD patients.

Due to the absence of multimodality imaging study in CAD patients, the investigators perform a large-scale, retrospective/prospective observational cohort study:

1. To identify the imaging and functional biomarkers related to CAD progression and clinical outcomes.
2. To evaluate the diagnostic and prognostic value of novel imaging biomarkers (CCTA pericoronary fat attenuation index, 18F-NaF PET/CT microcalcification, CMR T2 mapping, etc) for coronary and myocardial inflammation, and the association between novel imaging biomarkers and cerebral metabolism and inflammation
3. To evaluate the correlation and combination of different imaging/functional biomarkers (noninvasive or invasive) and develop the optimal imaging/functional biomarkers to predict recurrent CAD events.
4. To explore the effect of lifestyle or behaviors (eating habit, physical exercise, and sleeping pattern), social psychological and environmental factors on the occurrence, progression, and recurrence of CAD
5. To establish a novel risk stratification model including clinical factors, biomarkers and imaging markers, and explore the incremental predictive value of the novel model, in comparison to traditional clinical risk scores, for the prediction of clinical outcomes in CAD patients.

CCTA substudy: for patients with CCTA imaging, we aim to evaluate the diagnostic value and prognostic implication of one-stop CCTA test including degree of stenosis, lesions, CCTA-derived fractional flow reserve, shear force, and pericoronary adipose tissue, on culprit or high-risk lesions identified by optical coherence tomography (OCT).

PET-CT substudy: for patients with PET/CT examination, we aim to evaluate the association of neurometabolic activity by 18FDG PET/CT with plaque microcalcification by 18NaF PET/CT, pericoronary inflammation by CCTA, or high-risk plaque characteristics by OCT. Furthermore, the combined predictive value of these imaging markers will also be assessed.

CMR substudy: for STEMI patients with CMR, we aim to investigate the association of coronary angiography-derived index of microcirculatory resistance (angio-IMR) with myocardial injury and inflammation by CMR, and validate the prognostic value of combination of angio-IMR and CMR-derived parameters.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years old.
* 2. Patients with suspected or confirmed coronary artery disease who are eligible to undergo coronary angiography and IVUS/OCT or functional examination.
* 3. Written informed consent.
* 4. Subject is willing to comply with all protocol-required follow-up evaluation.

Exclusion Criteria:

* 1. Malignant tumor, lymphoma, HIV-positive, or cirrhosis with life expectancy <1 year.
* 2. Pregnancy, lactation, or potentially fertile women.
* 3. Patients who cannot complete this trial or comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected or confirmed CAD who are eligible to undergo coronary angiography and IVUS/OCT or functional tests.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-03-12 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events (MACEs) | Median 12 months
  Including cardiovascular death, nonfatal myocardial infarction, ischemia-driven revascularization

SECONDARY OUTCOMES:
Major adverse cardiac and cerebrovascular events (MACCEs) | Median 12 months
  Including cardiovascular death, nonfatal myocardial infarction, nonfatal stroke, ischemia-driven revascularization
Cardiovascular death | Median 12 months
All-cause death | Median 12 months
Myocardial infarction | Median 12 months
Stroke | Median 12 months
Heart failure | Median 12 months
Target vessel revascularization | Median 12 months
Revascularization | Median 12 months
Hospitalization for unstable angina | Median 12 months
Stent thrombosis | Median 12 months
Bleeding events (BARC 2,3,5) | Median 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Wang, MD, Principal Investigator — Beijing Anzhen Hospital
Locations (2):
- China (2):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No